CLINICAL TRIAL: NCT00430027
Title: Pilot Feasibility Trial of Preoperative Capecitabine, Oxaliplatin, Cetuximab and Radiation Therapy for Locally Advanced Esophageal Adenocarcinoma
Brief Title: Preoperative Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy for Locally Advanced Esophageal Adenocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due slow accrual.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0011.cc
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-10

CONDITIONS: Esophageal Adenocarcinoma
Keywords: Esophageal; Esophagus
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Capecitabine; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, oxaliplatin, cetuximab, and radiation therapy (Experimental): Patients enrolled on the trial will receive neoadjuvant combined capecitabine, oxaliplatin, cetuximab, and radiation therapy. This will be followed by surgical resection and adjuvant capecitabine, oxaliplatin, and cetuximab
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: Capecitabine — Given 650 mg/m^2 BID on days of ration therapy, 825 mg/m^2 day 1-14, day 15-20 off x 4
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin 30 mg/m^2, 130mg/m2 IV Q 21 days x 4
  Other Names: Eloxatin
Drug: Cetuximab — Initial Cetuximab 400 mg/m^2 IV starting no earlier than 8 weeks and no later than 10 weeks after surgical resection
  Other Names: Erbitux

SUMMARY:
The primary objective of this pilot study is to determine whether neoadjuvant capecitabine/oxaliplatin/cetuximab and external beam radiation therapy followed by surgical resection [and then followed by post operative adjuvant capecitabine, oxaliplatin and cetuximab] is feasible and tolerable.

DETAILED DESCRIPTION:
It is clear that new approaches are needed to improve the therapeutic ratio in esophageal cancer. This study proposes to evaluate the novel combination of preoperative capecitabine, oxaliplatin, and cetuximab concurrently with radiation therapy. This will be followed by esophagectomy 6-9 weeks after the completion of chemoradiation. Followed by further adjuvant chemotherapy. It is hypothesized that our novel combination of neoadjuvant capecitabine, oxaliplatin, and cetuximab combined with thoracoabdominal radiation therapy will be feasible and result in acceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients 18 years of age or older
* biopsy proven, non-recurrent primary adenocarcinoma of the thoracic esophagus or gastro-esophageal junction, disease confined to esophagus and peri-esophageal soft tissue, tumors at the gastroesophageal junction must be limited to no greater than 2 cm into the gastric cardia
* clinical stage T3, N0-1 or T1-2, N1 and M0 or M1a (celiac axis lymph nodes are allowed)
* Karnofsky Performance Status of >60%
* forced expiratory volume at one second (FeV1) must be >1.0 L
* adequate bone marrow reserve equal to or absolute neutrophil count (ANC) > 1500/mcl, total white blood cell count (WBC) > 3000/mcl, platelets >100,000/mcl and hemoglobin > 10.0 g/dl (transfusion permitted)
* adequate hepatic function of direct serum bilirubin < 2 times the upper limit of normal, total bilirubin < 1.5 times the upper limit normal, alanine transaminase (ALT), aspartate transaminase (AST) < 2.5 times the upper limit normal, Alkaline phosphatase < 2.5 times the upper limit normal
* creatinine clearance > 50 ml/min
* female patients of childbearing potential must have a negative serum or urin pregnancy test within 7 days prior to starting therapy

Exclusion Criteria:

* no previous resection or attempted resection of an esophageal cancer
* women who are pregnant or lactating
* life expectancy < 3 months
* serious, uncontrolled concurrent infection(s)
* prior fluoropyrimidine therapy
* prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil or known Dihydro Pyrimidine Dehydrogenase Deficiency (DPD) deficiency
* treatment for other carcinomas within 5 years, except cured non-melanoma skin and treated in-situ cervical cancer
* history of or evidence of uncontrolled diabetes
* surgical procedure within 6 months of study entry
* participation in any investigational drug study within 4 weeks preceding the start of study treatment
* prior therapy with andy agent that specifically targets the Epidermal Growth Factor Receptor (EGFR) pathway
* prior severe infusion reaction to a monoclonal antibody
* acute hepatitis or known HIV
* clinically significant cardia disease
* evidence of metastases
* other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* major surgery within 4 weeks of the start of treatment without complete recovery
* lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* known, existing uncontrolled coagulopathy
* unwillingness to give written informed consent
* unwillingness to participate or inability to comply with the protocol for the duration of the study
* neuropathy of grade 2 or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Schefter, MD, Principal Investigator — University of Colorado at Denver and Health Science Center
Locations (1):
- University of Colorado at Denver and Health Science Center, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2006 and August 2008, 8 patients were enrolled in the study from the Radiation Oncology clinic.
Pre-assignment Details: This was to be a pilot/feasibility trial with a maximum of 15 patients enrolled, with the intent to propose a phase II trial. The study stopped before enrolling 15 patients, therefore the phase II trial was not pursued.
Groups:
- Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy: Patients enrolled on the trial received neoadjuvant combined capecitabine, oxaliplatin, cetuximab, and radiation therapy. This was followed by surgical resection and adjuvant capecitabine, oxaliplatin, and cetuximab
Period: Overall Study
Arm/Group | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study terminated | 8

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Toxicity
Description: The primary objective of this pilot study was to determine whether neoadjuvant capecitabine/oxaliplatin/cetuximab and external beam radiation therapy followed by surgical resection and then followed by post operative adjuvant capecitabine, oxaliplatin and cetuximab is feasible with acceptable toxicity profile.
Time Frame: Up to 4 weeks
Population: The study was terminated, study end points were not reached.
Arm/Group | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for approximately 2 years.
Description: Patients were assessed weekly at their clinic visits.
Arm/Group | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy (N=8)
Infection (Infections and infestations) | 1 (1) — Septic shock
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Cetuximab, and Radiation Therapy (N=8)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Distension (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 6 (21)
INR (Investigations) | 3 (11)
Hypersensitivity (Immune system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1) — Abdominal cramping
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Pericardial effusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated due slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes